CLINICAL TRIAL: NCT00864942
Title: Phase I Clinical Trial of Bendamustine, Lenalidomide and Rituximab in B-Cell Lymphoid Malignancies
Brief Title: Trial of Bendamustine, Lenalidomide and Rituximab in Chronic Lymphocytic Leukemia (CLL) and Non-Hodgkin's Lymphoma (NHL)
Acronym: Phase I BLR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Celgene Corporation (Industry); Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RV-CLL-NHL-PI-356; 2008-186
Record Dates: First submitted 2009-03-17; First posted 2009-03-19 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Lymphocytic Leukemia; Non-Hodgkin's Lymphoma
Keywords: CLL; NHL; lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin; Lymphoma | interventions — Bendamustine Hydrochloride; Lenalidomide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- BL-NHL (Experimental): Bendamustine and lenalidomide for NHL
  Interventions: Drug: BL-NHL
- BLR-CLL (Experimental): Bendamustine, lenalidomide, rituximab for CLL
  Interventions: Drug: BLR-CLL
- BLR-NHL (Experimental): Bendamustine, lenalidomide, and rituximab for NHL
  Interventions: Drug: BLR-NHL
- BL-CLL (Experimental): bendamustine and lenalidomide in patients with CLL
  Interventions: Drug: bendamustine and lenalidomide

INTERVENTIONS:
Drug: bendamustine and lenalidomide — Lenalidomide is given daily orally for one week followed by bendamustine HCL 90 mg/m2 IV over 30 to 60 minutes on days 1 and 2 in combination with lenalidomide, given orally, in dose-escalating cohorts. After a maximum of 6 cycles of combination therapy with bendamustine and lenalidomide, lenalidomide monotherapy is continued for an additional 6 cycles as tolerated or until disease progression.
  Other Names: Bendamustine HCL; Treanda; Revlimid
  Arms: BL-CLL
Drug: BL-NHL — Bendamustine HCL 90 mg/m2 given intravenously over 30 to 60 minutes on days 1 and 2 in combination with lenalidomide, given orally, in dose-escalating cohorts. After a maximum of 6 cycles of combination therapy with bendamustine and lenalidomide, lenalidomide monotherapy is continued for an additional 6 cycles as tolerated or until disease progression.
  Other Names: Bendamustine HCL; Treanda; Revlimid
  Arms: BL-NHL
Drug: BLR-CLL — Lenalidomide is given orally for 7 days followed by rituximab 375 mg/m2 on day 1 in addition to bendamustine 90 mg/m2 intravenously over 30-60 minutes on days 1 and 2 and lenalidomide orally daily every 28 days for a total of 6 cycles. After 6 cycles of bendamustine, lenalidomide and rituximab, lenalidomide monotherapy is administered as continued therapy for an additional 6 cycles as tolerated or until disease progression.
  Other Names: Bendamustine HCL; Treanda; Revlimid; Rituxan
  Arms: BLR-CLL
Drug: BLR-NHL — Rituximab 375 mg/m2 is given on day 1 on day 1 in addition to bendamustine 90 mg/m2 intravenously over 30-60 minutes on days 1 and 2 and lenalidomide orally daily every 28 days for a total of 6 cycles. After 6 cycles of bendamustine, lenalidomide and rituximab, lenalidomide monotherapy is administered as continued therapy for an additional 6 cycles as tolerated or until disease progression.
  Other Names: Bendamustine HCL; Treanda; Revlimid; Rituxan
  Arms: BLR-NHL

SUMMARY:
This study is for subjects with a B-cell lymphoid malignancy (lymphoma) or chronic lymphocytic leukemia (CLL) that has come back after or did not get better with previous treatment. The purpose of this study is to find out the highest dose of lenalidomide that can be given together with bendamustine and rituximab. The study will also look what effects the combination of lenalidomide and bendamustine and the combination of lenalidomide, bendamustine and rituximab will have on patients and their disease.

DETAILED DESCRIPTION:
This is a Phase I, open-label, dose-escalation study of bendamustine and lenalidomide (BL) and also bendamustine,lenalidomide, and rituximab (BLR) in relapsed/refractory CLL and relapsed/refractory B-cell lymphomas. Phase I dose escalation will be done independently for the CLL and NHL groups. In addition, the study will be conducted in 2 parts. In part I of the study, the maximum tolerated dose of bendamustine and lenalidomide will be determined independently for the CLL and NHL groups. In part II of the study, CLL and NHL subjects will be enrolled at the MTD of BL determined in Part I for CLL and NHL and all subjects will receive rituximab. Part II of the study will determine the MTD of BLT independently for the NHL and CLL groups.

ELIGIBILITY:
Inclusion Criteria:

* Documented relapsed or refractory B-cell NHL; CD-20 positive tumor. Indolent NHL: follicular B-cell lymphoma, diffuse small lymphocytic lymphoma, lymphoplasmacytic lymphoma, marginal zone lymphoma, transformed aggressive lymphomas, mantle cell lymphoma and chronic lymphocytic leukemia
* Maximum of 6 prior chemotherapy regimens. Prior rituximab is allowed.
* Bidimensionally measurable disease
* ECOG performance status 0-2
* Absolute neutrophil count >/= 1000 and platelet count >/= 50,000
* Serum creatinine </= 1.5 mg/dL
* Adequate hepatic function
* Estimated life expectancy of at least 3 months
* All study participants must be registered into the mandatory RevAssist program and be willing and able to comply with the requirements of RevAssist
* Able to take aspirin 81 mg daily as prophylactic anticoagulation

Exclusion Criteria:

* Chemotherapy or immunotherapy within 3 weeks prior to entering study or failure to recover from adverse events due to any agents administered previously
* Use of investigational agents within 28 days of study
* Hematopoietic growth factors within 14 days of study
* History of prior high dose chemotherapy with allogeneic stem cell support
* History of prior radioimmunotherapy </= 1 year
* Concurrent treatment with therapeutic doses of systemic steroids
* Pregnant or lactating female subjects
* Concurrent, active malignancy other than lymphoma or CLL
* Primary CNS lymphoma
* Patients with a prior diagnosis of lymphoma active in the CNS are eligible only if CNS has been treated, and they are neurologically stable with no progressive symptoms off steroids and anti-convulsants
* Serious infection, medical condition, or psychiatric condition that, in the opinion of the investigator, might interfere with the achievement of study objectives
* Hypersensitivity to murine proteins or to any component of rituximab
* Known positive for HIV or infectious hepatitis type C; hepatitis type B that is active and uncontrolled
* Hypersensitivity to mannitol
* Evidence of laboratory tumor lysis syndrome by Cairo-Bishop criteria
* Subject with recent thromboembolic event (deep vein thrombosis or pulmonary embolism) unless clinically stable and event occurred more than 2 weeks prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 2 years
Dose limiting toxicity | 2 years
Recommended Phase II dose | 2 years

SECONDARY OUTCOMES:
overall safety profile | 2 years
Plasma pharmacokinetics | 2 years
Preliminary antitumor activity | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bruce D Cheson, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University Hospital/Lombardi Cancer Center, Washington D.C., District of Columbia, United States